CLINICAL TRIAL: NCT00620724
Title: Maintenance Oral Nifedipine for Management of Symptomatic Placenta Previa : A Randomized Clinical Trial
Brief Title: Tocolytic Therapy in Conservative Management of Symptomatic Placenta Previa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005/065/HP
Record Dates: First submitted 2008-01-28; First posted 2008-02-21 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Placebo Comparator): Placebo three times daily
  Interventions: Drug: Placebo
- B (Experimental): 20 mg of slow-release Nifedipine three times daily
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Placebo — Placebo three times daily
  Arms: A
Drug: Nifedipine — 20 mg of slow-release Nifedipine three times daily
  Arms: B

SUMMARY:
The objective of our study is to determine the clinical utility related to the maintenance oral nifedipine therapy in patients with symptomatic placenta previa. This study is a prospective, randomized controlled trial with the inclusion, after 24 weeks gestation, of hospitalized patients with symptomatic placenta praevia. All patients may initially receive oral nifedipine therapy with steroid prophylaxis for 48 hours. After then, patients are randomly assigned to receive either oral nifedipine (20 mg every 8 hours) or placebo (one every 8 hours) until 37 weeks of gestation.

The primary outcome for the trial is the length of pregnancy in days after the enrollment. A sample size calculation is designed to detect at least a 14 -day difference in time gained in patients with maintenance oral nifedipine therapy. A sample size of about 52 patients per group would have a 80 % chance of detecting this difference at the 5 % level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Placenta previa is diagnosed when the lowest placental edge is located within 5 cm of the internal os at ultrasonography
* Placenta previa may be symptomatic with at least one episode of bleeding
* Estimated gestational age within 24 to 34 weeks
* Maternal age > 18 years
* Informed consent after received an explanation of the study and an information sheet
* Social affiliation

Exclusion Criteria:

* Premature rupture of membranes
* Severe bleeding requiring an immediate termination of pregnancy
* Abnormal fetal heart rates requiring an immediate termination of pregnancy
* Intrauterine fetal death
* Pre-eclampsia, chorioamnionitis, liver disease, severe chronic renal disease, heart disease
* Abruptio placentae
* Nifedipine sensibility
* Drugs interaction with nifedipine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-01; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Prolongation of pregnancy | From allocation to the delivery

SECONDARY OUTCOMES:
Maternal outcomes i.e number episodes of bleeding, amount of bleeding, number of blood transfusion required | At the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Rouen, Rouen, France

REFERENCES:
- [Derived] Verspyck E, Thill C, Ego A, Machevin E, Brasseur-Daudruy M, Ickowicz V, Blondel C, Degre S, Lefebure A, Braund S, Benichou J. Screening for small for gestational age infants in early vs late third-trimester ultrasonography: a randomized trial. Am J Obstet Gynecol MFM. 2023 Nov;5(11):101162. doi: 10.1016/j.ajogmf.2023.101162. Epub 2023 Sep 15. PMID 37717697
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046
- [Derived] Verspyck E, de Vienne C, Muszynski C, Bubenheim M, Chanavaz-Lacheray I, Dreyfus M, Deruelle P, Benichou J. Maintenance nifedipine therapy for preterm symptomatic placenta previa: A randomized, multicenter, double-blind, placebo-controlled trial. PLoS One. 2017 Mar 23;12(3):e0173717. doi: 10.1371/journal.pone.0173717. eCollection 2017. PMID 28333939